CLINICAL TRIAL: NCT06012526
Title: Study of the Prevalence and Predictive Factors of Sleep Disordered Breathing in Patients With Interstitial Lung Diseases
Brief Title: The Study of Sleep Disordered Breathing in Patients With Interstitial Lung Diseases
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mona Mahmoud Srour Soliman, Assistant lecturer, Beni-Suef University
Other Study IDs: BeniSuefU MMSS
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Obstructive Sleep Apnea-hypopnea
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA group: The group of patients who had sleep disordered breathing
  Interventions: Diagnostic Test: Polysomnography
- No OSA group: The group of patients who had not sleep disordered breathing
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Polysomnography is done for patients to find any sleep disordered breathing
  Other Names: Sleep study

SUMMARY:
This was a cross-sectional observational study to evaluate the prevalence and predictive factors of SDB in ILD and to analyze the relationship between polysomnography (PSG) findings, pulmonary function, disease severity, parenchymal involvement, and sleep questionnaires ESS and SBQ. This study included 69 patients who were diagnosed with diffuse parenchymal lung diseases by high-resolution computed tomography (HRCT) chest. All patients were subjected to clinical examination, HRCT, spirometry, full-night polysomnography, and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes of clinically stable ILD patients older than 18 who met the ATS/ERS criteria for an ILD diagnosis were included in the study.

Exclusion Criteria:

* Patients who have any anatomic upper airway obstructions such as significant nasal septal deviation, nasal polyps, conchae hypertrophy or tonsillar hypertrophy.
* Patients with neurological diseases or severe psychiatric disorders.
* Patients who have history of administration of any drug that has a major effect on sleep e.g. benzodiazepine, narcotic drugs ….etc.
* Patients with any chronic pulmonary disease except ILD.
* Total sleep time less than 4 hours on PSG.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 69 patients with interstitial lung diseases of both sexs and older than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
Measurements of apnea hypopnea index | 1and half years
  Polysomnography can measure apnea hypopnea index of all patients to detect sleep disordered breathing

CONTACTS AND LOCATIONS:
Overall Officials: Nabila Ebrahim Laz, Professor, Study Chair — Head of chest department in BeniSuef university
Locations (1):
- Beni suef university, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
E mail address only can be shared
Supporting Information: Study Protocol, SAP